CLINICAL TRIAL: NCT07283458
Title: TICOALA-SOINS : Assessment of Language Comprehension and Learning in Children Attending Child Psychiatry Services. Pilot Study of Acceptability and Feasibility.
Brief Title: Assessment of Language Comprehension and Learning in Children Attending Child Psychiatry Services (TICOALA-SOINS)
Acronym: TICOALA-SOINS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Université Paris Cité (Other); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D25-P001
Record Dates: First submitted 2025-11-20; First posted 2025-12-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Typical Development; Typically Developing Children Ages 3 to 6; Typical Preschoolers Who Can Not Zipper; Children; Children Behavior Problem; FRENCH STUDY
Keywords: language assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with language comprehension and learning difficulties (Other)
  Interventions: Other: TICOALA

INTERVENTIONS:
Other: TICOALA — The TICOALA tool (Interactive Test of Language Comprehension and Learning on tablet) offers a quick and engaging way to evaluate children's lexical and syntactic comprehension, as well as their ability to learn new words. Integrating this tool into clinical practice could provide an initial language assessment and help guide referrals for formal speech-language evaluation.

SUMMARY:
Language is central to children's cognitive, emotional, and social development, and language difficulties are a frequent reason for consultation in child psychiatry, often co-occurring with psychiatric disorders. Yet, systematic language assessment is rarely possible due to the limited availability of speech-language therapists in these services.

The TICOALA tool (Interactive Test of Language Comprehension and Learning on tablet) offers a quick and engaging way to evaluate lexical and syntactic comprehension and word learning. This study aims to assess its acceptability among children aged 3-7 attending a child psychiatry service in Paris, as well as among clinicians and parents. Secondary goals include testing the feasibility of a larger study, describing children's language skills, and examining how these relate to clinical and background variables.

DETAILED DESCRIPTION:
Language is intrinsically linked to children's cognitive, social, emotional, and psychological development, and plays a crucial role in both academic achievement and psychosocial adjustment. In child psychiatry, language difficulties are a common reason for consultation and are frequently associated with psychiatric conditions such as anxiety disorders or attention difficulties. However, due to the limited availability of speech-language therapists in these settings, systematic language assessments are rarely conducted.

The TICOALA tool (Interactive Test of Language Comprehension and Learning on tablet) offers a quick and engaging way to evaluate children's lexical and syntactic comprehension, as well as their ability to learn new words. Integrating this tool into clinical practice could provide an initial language assessment and help guide referrals for formal speech-language evaluation.

Main Objective To assess the acceptability of the TICOALA tool among children attending our child psychiatry service.

Secondary Objectives

* To evaluate its acceptability for clinicians (psychiatrists, psychologists) and parents.
* To assess the acceptability of the parental clinical questionnaire.
* To determine the feasibility of conducting a larger-scale study.
* To describe the language skills (lexical, syntactic, word learning) of children in our service.
* To analyze the relationship between language skills and clinical/anamnestic data (socio-economic background, play and screen exposure, language experience, etc.).

Target Population Children aged 3-7 years consulting at the child psychiatry service in the 14th arrondissement of Paris.

ELIGIBILITY:
Inclusion Criteria:

* Children (boys or girls) aged 3-7 years
* Consulting in the child psychiatry service
* Enrolled in a French-speaking school

Exclusion Criteria:

* Inability to use the tablet-based TICOALA tool due to severe sensory (blindness, deafness), motor, or intellectual impairment
* Refusal of the child or parents/legal guardians to participate
* Child not affiliated with the French social security system

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2028-03-03 (Estimated); Study Completion 2028-03-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the TICOALA tool among children attending our child psychiatry service | 4 months
  This objective will be evaluated using a questionnaire with a 5-point Likert scale, with a composite evaluation criterion based on three elements: the child's opinion, their level of attention, and their level of motivation. The questionnaire will be completed by the consultant, reporting the child's opinion and their clinical observations (attention, motivation) during the assessment.

IPD SHARING:
Plan to Share IPD: Yes
Only anonimyzed results will be shared. Each child will be assigned a code. Data shared will simply include scores on the tasks and answers in the questionnaires without any information linked to each individual identity.
Supporting Information: Study Protocol, SAP, Analytic Code